CLINICAL TRIAL: NCT00004482
Title: Phase II Randomized Study of Muromonab-CD3, Cyclosporine, Methylprednisolone, and Prednisone in Patients With Giant Cell Myocarditis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/14209; MAYOC-1479901; MAYOC-1479900
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Myocarditis; Giant Cell Myocarditis
Keywords: cardiovascular and respiratory diseases; giant cell myocarditis; rare disease
MeSH Terms: conditions — Myocarditis; Respiratory Tract Diseases; Rare Diseases | interventions — Cyclosporine; Methylprednisolone; Muromonab-CD3; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cyclosporine
Drug: methylprednisolone
Drug: Muromonab-CD3
Drug: prednisone

SUMMARY:
OBJECTIVES:

I. Assess the effect of immunosuppression with muromonab-CD3, cyclosporine, methylprednisolone, and prednisone versus standard care in terms of death, heart transplantation, or left ventricular assistive device placement in patients with giant cell myocarditis.

II. Compare left ventricular ejection fraction prior to and after 4 weeks of treatment in these arms.

III. Compare the degree of myocardial inflammatory infiltrate prior to and after 4 weeks of treatment in these arms.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, open label, multicenter study.

Patients are randomized to receive standard care with immunosuppression (arm I) or standard care with or without immunosuppression (no muromonab-CD3 or cyclosporine)(arm II).

Arm I: Patients receive methylprednisolone IV once daily for 3 days and muromonab-CD3 IV once daily for 10 days. Oral cyclosporine is administered twice daily and oral prednisone is administered once daily for 1 year.

Arm II: Patients receive standard care with or without immunosuppression (no muromonab-CD3 or cyclosporine).

Patients are followed for one year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Idiopathic giant cell myocarditis confirmed by endomyocardial biopsy

Heart failure and/or arrhythmia of less than 3 months duration

--Patient Characteristics--

Hepatic: AST/ALT no greater than 3 times upper limit of normal

Renal: Creatinine no greater than 2.5 mg/dL

Other: Not pregnant or nursing; Negative pregnancy test; Fertile patients must use effective contraception; No clinical evidence of sepsis or active infection (e.g. meningitis, osteomyelitis, etc.); No contraindication to immunosuppression; No allergy to cyclosporine or muromonab-CD3; No other severe concurrent diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1999-12; Primary Completion 2005-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie T. Cooper, Jr., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States